CLINICAL TRIAL: NCT01158378
Title: A Pivotal Clinical Trial Examining the Safety and Effectiveness of the Adherus Dural Sealant System When Used as a Dural Sealant in Cranial Procedures
Brief Title: Safety and Effectiveness of the Adherus Dural Sealant System When Used as a Dural Sealant in Cranial Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HyperBranch Medical Technology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HBMT-080453
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-02

CONDITIONS: Elective Cranial Procedures With Dural Incision
Keywords: Adherus Dural Sealant; Adherus AutoSpray Dural Sealant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DuraSeal Dural Sealant System (Active Comparator)
  Interventions: Device: Adherus Dural Sealant
- Adherus Dural Sealant System (Experimental)
  Interventions: Device: Adherus Dural Sealant

INTERVENTIONS:
Device: Adherus Dural Sealant — In situ polymerizing sealant

SUMMARY:
The purpose of the study is to demonstrate the safety and effectiveness of the Adherus Dural Sealant System when used as a dural sealant in conjunction with standard methods of dural repair in cranial procedures.

DETAILED DESCRIPTION:
After surgery on the head, the dura, a membrane that covers the brain, must be closed in order to prevent CSF from leaking outside of the dura. When CSF leaks outside the dura, this can increase the risk of infection, cause painful headaches or complications that may require another surgery to repair the leak. Typically, your study doctor will close the dura with sutures (surgical stitches) and sometimes a piece of muscle, fat, or other soft tissue taken from another place on your body. However, it is still possible that CSF will continue to leak through small suture holes even when all appropriate precautions have been taken.

Dural surgical sealants have been developed to assist surgeons in stopping CSF leaks when standard measures following brain surgery are not effective. Sometimes, the leak seals on its own and there is no need for a surgical sealant.

This study is for participants who have a CSF leak after standard measures are used to close the dura at the end of their surgery. The decision to use a surgical sealant will be made when your surgeon finds that after stitching and using standard measures to close the dura, there is still a leak.

However, if your surgeon finds a CSF leak after he or she applies the standard stitches and tissues, and you have signed this informed consent, then you will be randomized to receive one of two surgical sealants (Randomized means like a flip of the coin). You will be selected to receive either Adherus™ Surgical Sealant or DuraSeal™ Surgical Sealant and your post surgery progress will be evaluated during study visits and with study tests. Adherus™ Surgical Sealant is an investigational device that has been developed to stop CSF leaks. It is being studied to find if it is just as effective and safe as DuraSeal™.

Adherus™ is made of two components that form a gel when they are combined. The gel is applied after the study doctor closes the incision. The gel acts as a thin, elastic barrier intended to prevent CSF from leaking until the dura tissue has properly healed on its own. The gel is then absorbed by the body over several months and excreted or removed from the body through the urine. This is the second study of Adherus™ in people in the United States.

If you choose to participate, you will have screening tests to see if you qualify to enroll in the study. Not everyone who is screened for the study will be able to participate. The device you receive will be determined by a random selection process. Neither you nor study personnel or your doctor can decide which device you receive. You will not be told which device you received until study completion. In addition, if your study doctor does not use any sealant at the end of your surgery (you may not have any CSF leak or the study doctor decides to use another closure procedure) then your study participation will be complete.

If you choose to participate and have screening tests to qualify you to enroll in the study, your surgery will be performed according to the regular standard of care. If CSF leaks from your dura after it is stitched closed by your study doctor and you continue to meet study entry measures, then your study doctor will apply the assigned study treatment to try to stop the leak. After the surgery, you will be seen 4 times over the next 4 months. You will be in the study for up to 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Pre-Operative Inclusion Criteria
* Subject is scheduled for an elective cranial procedure involving a dural incision using any of the following surgical locations/approaches (or combination): frontal, temporal, occipital, and parietal (i.e. supratentorial), and/or midline or lateral suboccipital (i.e. infratentorial.) Subject requires a procedure involving a Class 1/clean wound (uninfected surgical wound in which no inflammation is encountered)

Intra-Operative Inclusion Criteria

* Subject's linear extent of durotomy is ≥2 cm
* Subject's dural margins from the edges of bony defect are ≥3 mm throughout
* Subject's CSF leak is present intra-operatively following completion of primary dural closure (with or without non-autologous duraplasty or autologous tissue), either spontaneously or upon Valsalva maneuver, at up to 20 cm H2O for up to five (5) seconds

Exclusion Criteria:

* Subject requires a procedure involving a translabyrinthine, transsphenoidal, transoral approach, or any procedure that penetrates the air sinus or mastoid air cells. Note: Superficial penetration of mastoid air cells is not an exclusion if cells are appropriately sealed (e.g. bone wax).
* Subject has a CSF shunt such as; ventriculo-peritoneal, ventriculo-pleural, ventriculo-atrial or lumbo-peritoneal shunts.
* Subject has an external ventricular or lumbar CSF drain that must be left in place after surgery.
* Subject has had radiation treatment to the surgical site, or standard fractionated radiation therapy is planned within ten days post index-procedure. (Note: stereotactic radiosurgery prior to the planned index procedure is not an exclusion criterion).
* Subject has a systemic infection or evidence of any infection near planned operative site.

Intra-Operative Exclusion Criteria

* Subject has an Incidental finding that meets any pre-operative exclusion criterion listed above.
* Subject requires the intra-operative placement of a CSF diversion device (e.g. ventricular catheter, subdural catheter, lumbar drain, or other device designed to externally evacuate CSF) that will be left in place after the procedure. Note: Subgaleal drains used for acute post-operative management of the incision site are permitted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Smith, MD, Principal Investigator — Carolina Neurosurgery & Spine Associates
Locations (17):
- United States (17):
  - Colorado Brain and Spine Institute/Swedish Medical Center, Englewood, Colorado
  - Florida Hospital, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Wayne State University, Detroit, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - Saint Louis University, St Louis, Missouri
  - Stony Brook University Medical Center, Stony Brook, New York
  - Carolina Neurosurgery & Spine Associates, Charlotte, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Mayfield Clinic, Cincinnati, Ohio
  - Oklahoma Spine and Brain Institute, Tulsa, Oklahoma
  - Penn State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Background] Bakar B, Kose EA, Balci M, Atasoy P, Sarkarati B, Alhan A, Kilinc K, Keskil IS. Evaluation of the neurotoxicity of the polyethylene glycol hydrogel dural sealant. Turk Neurosurg. 2013;23(1):16-24. doi: 10.5137/1019-5149.JTN.6039-12.1. PMID 23344862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was treated on September 3, 2010 and the last subject visit occurred on January 17, 2013.
Pre-assignment Details: Randomized study, no washout or run-in period.
Groups:
- DuraSeal Dural Sealant System: DuraSeal Dural Sealant System: In situ polymerizing sealant
Period: Overall Study
Arm/Group | Adherus Dural Sealant | DuraSeal Dural Sealant System
Started | 124 | 126
Completed | 114 | 117
Not Completed | 10 | 9
Not completed — Death | 4 | 5
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Population: Only subjects with unknown cranial endpoint status, who died of known causes unrelated to the study device or procedure were excluded from baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adherus Dural Sealant | DuraSeal Dural Sealant System | Total
Number analyzed (Participants) | 120 | 122 | 242
Age, Customized [Mean (Standard Deviation); unit: years] | 51.1 (14.0) | 49.6 (15.1) | 50.4 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 79 | 84 | 163
Region of Enrollment [Number; unit: participants]
  United States | 120 | 122 | 242

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Treated Subjects Who Were Free of Intra-operative Cerebrospinal Fluid (CSF) Leakage From Dural Repair During Valsalva Maneuver, CSF Leak / Pseudomeningocele, and Unplanned Retreatment of the Original Surgical Site
Description: The primary endpoint was a composite evaluation of the safety and effectiveness of Adherus for a cranial application. The endpoint was measured by the proportion of treated subjects who were free of all of the following incidences:
  * Intra-operative CSF leakage from dural repair after up to two Adherus / control applications during Valsalva maneuver up to 20cm H2O for up to 5 seconds.
  * CSF leak or pseudomeningocele diagnosed by physical examination, biochemical assay or imaging study during the 120-day follow-up period of the index procedure
  * Unplanned retreatment of the original surgical site adjudicated by the CEC to be device-related, including meningitis or the management of deep infection, minimally invasive procedures or return to the operating room for neurosurgical complications other than CSF leak or pseudomeningocele formation or those related to the subject's pre-existing condition, during the 120-day follow-up period.
Time Frame: 120 days
Population: All subjects who received treatment with evaluable 120-day follow-up data.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Adherus Dural Sealant System | DuraSeal Dural Sealant System
Number analyzed (Participants) | 114 | 117
percentage of subjects | 91.2 [84.5 to 95.7] | 90.6 [83.8 to 95.2]
Statistical Analysis 1: Comparison: Adherus Dural Sealant System vs DuraSeal Dural Sealant System; Test type: Non-Inferiority or Equivalence — non-inferiority margin of 10%; p = 0.0049, one-sided z-test

2. Post Hoc Outcome: Proportion of Treated Subjects Who Were Free of Intra-operative Cerebrospinal Fluid (CSF) Leakage From Dural Repair During Valsalva Maneuver, CSF Leak / Pseudomeningocele, and Unplanned Retreatment of the Original Surgical Site
Description: Post-Hoc analysis of primary composite endpoint of the safety and effectiveness of Adherus for a cranial application at 14 days. The endpoint was measured by the proportion of treated subjects who were free of all of the following incidences:
  * Intra-operative CSF leakage from dural repair after up to two Adherus / control applications during Valsalva maneuver up to 20cm H2O for up to 5 seconds.
  * CSF leak or pseudomeningocele diagnosed by physical examination, biochemical assay or imaging study during the 120-day follow-up period of the index procedure
  * Unplanned retreatment of the original surgical site adjudicated by the CEC to be device-related, including meningitis or the management of deep infection, minimally invasive procedures or return to the operating room for neurosurgical complications other than CSF leak or pseudomeningocele formation or those related to the subject's pre-existing condition, during the 120-day follow-up period.
Time Frame: 14 days
Population: All subjects who received treatment with evaluable 14-day follow-up data.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Adherus Dural Sealant System | DuraSeal Dural Sealant System
Number analyzed (Participants) | 117 | 120
percentage of subjects | 99.1 [95.3 to 100] | 95.0 [89.4 to 98.1]
Statistical Analysis 1: Comparison: Adherus Dural Sealant System vs DuraSeal Dural Sealant System; Test type: Non-Inferiority or Equivalence — non-inferiority margin of 10%; p < 0.0001, one-sided z-test
Statistical Analysis 2: Comparison: Adherus Dural Sealant System vs DuraSeal Dural Sealant System; Superiority Test; Test type: Superiority or Other; p = 0.0297, one-sided z-test

3. Post Hoc Outcome: Proportion of Treated Subjects Who Were Free of Intra-operative Cerebrospinal Fluid (CSF) Leakage From Dural Repair During Valsalva Maneuver, CSF Leak / Pseudomeningocele, and Unplanned Retreatment of the Original Surgical Site
Description: Post-Hoc analysis of primary composite endpoint of the safety and effectiveness of Adherus for a cranial application at 45 days. The endpoint was measured by the proportion of treated subjects who were free of all of the following incidences:
  * Intra-operative CSF leakage from dural repair after up to two Adherus / control applications during Valsalva maneuver up to 20cm H2O for up to 5 seconds.
  * CSF leak or pseudomeningocele diagnosed by physical examination, biochemical assay or imaging study during the 120-day follow-up period of the index procedure
  * Unplanned retreatment of the original surgical site adjudicated by the CEC to be device-related, including meningitis or the management of deep infection, minimally invasive procedures or return to the operating room for neurosurgical complications other than CSF leak or pseudomeningocele formation or those related to the subject's pre-existing condition, during the 120-day follow-up period.
Time Frame: 45 days
Population: All subjects who received treatment with evaluable 45-day follow-up data.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Adherus Dural Sealant System | DuraSeal Dural Sealant System
Number analyzed (Participants) | 119 | 123
percentage of subjects | 96.6 [91.6 to 99.1] | 91.9 [85.6 to 96.0]
Statistical Analysis 1: Comparison: Adherus Dural Sealant System vs DuraSeal Dural Sealant System; Test type: Non-Inferiority or Equivalence — non-inferiority margin of 10%; p < 0.0001, one-sided z-test
Statistical Analysis 2: Comparison: Adherus Dural Sealant System vs DuraSeal Dural Sealant System; Superiority Test; Test type: Superiority or Other; p = 0.0561, one-sided z-test

4. Secondary Outcome: Proportion of Subjects Free of Device-related Surgical Wound Infections or Meningitis During 120-day Follow-up.
Description: Device-related surgical wound infections included all infections classified by the CEC as definitely, probably, possibly or undetermined in relation to the device.
Time Frame: 120 days
Population: Includes all subjects with available data that through 120 days follow-up.
Measure: Number; unit: percentage of subjects
Arm/Group | Adherus Dural Sealant | DuraSeal Dural Sealant System
Number analyzed (Participants) | 114 | 117
percentage of subjects | 100 | 98.3

ADVERSE EVENTS:
Time Frame: 120 days
Arm/Group | Adherus Dural Sealant System | DuraSeal Dural Sealant System
Serious Adverse Events (participants affected / at risk) | 33/124 | 33/126
Other Adverse Events (participants affected / at risk) | 28/124 | 29/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adherus Dural Sealant System (N=124) | DuraSeal Dural Sealant System (N=126)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Deafness Unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diverticular Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse Drug Reaction (General disorders) | 0 (0) | 2 (2)
Disease Progression (General disorders) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Incision Site Infection (Infections and infestations) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Brain Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain Herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pseudomeningocele (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Radiation Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal Ganglia Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrospinal Fluid Rhinorrhoea (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 3 (3)
Convulsion (Nervous system disorders) | 3 (3) | 0 (0)
Dyspraxia (Nervous system disorders) | 1 (1) | 0 (0)
Embolic Stroke (Nervous system disorders) | 2 (2) | 1 (1)
Gran Mal Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial Hypotension (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial Venous Sinus Thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Thalamic Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
VIIth Nerve Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Vocal Cord Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Panic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Drug Rash With Eosinophilia and Systemic Symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adherus Dural Sealant System (N=124) | DuraSeal Dural Sealant System (N=126)
Vision Blurred (Eye disorders) | 7 (7) | 7 (7)
Dizziness (Nervous system disorders) | 7 (7) | 4 (4)
Headache (Nervous system disorders) | 13 (14) | 16 (17)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No